CLINICAL TRIAL: NCT03392038
Title: Root Coverage Using the Coronally Positioned Tunnel Technique Comparing Thick Versus Thin Acellular Dermal Matrix
Brief Title: Thick vs. Thin Acellular Dermal Matrix (ADM)
Acronym: ADM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Louisville (Other)
Responsible Party: Principal Investigator, Henry Greenwell, Director, Graduate Periodontics, University of Louisville
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 16.0462
Record Dates: First submitted 2017-12-31; First posted 2018-01-05 (Actual); Last update posted 2020-09-10 (Actual); Status verified 2020-09

CONDITIONS: Gingival Recession
MeSH Terms: conditions — Gingival Recession

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Thin ADM (Experimental): Periodontal root coverage surgery using a coronally positioned tunnel and thin acellular dermal matrix (ADM GBR)
  Interventions: Procedure: Thin ADM
- Thick ADM (Active Comparator): Periodontal root coverage surgery using coronally positioned tunnel surgery and thick acellular dermal matrix graft (ADM)
  Interventions: Procedure: Thick ADM

INTERVENTIONS:
Procedure: Thin ADM — Use of soft tissue allograft for root coverage
  Other Names: Thin acellular dermal matrix (ADM GBR)
  Arms: Thin ADM
Procedure: Thick ADM — Periodontal surgical procedure to coronally position the tissue over the ADM allograft
  Other Names: Thick acellular dermal matrix graft (ADM)
  Arms: Thick ADM

SUMMARY:
To study and compare a thick vs thin acellular dermal matrix for root coverage using the coronally positioned tunnel technique.

ELIGIBILITY:
Inclusion Criteria:

A. At least one Miller Class I or II mucogingival defect ≥ 3 mm (Miller 1985). B. The mucogingival defect must be on a non-molar tooth. C. Patients must be ≥ 18 years of age.

Exclusion Criteria:

A. Patients with debilitating systemic or diseases that significantly affect the periodontium.

B. Patients with a known allergy to any of the materials that will be used in the study, including systemic antibiotics (tetracycline and doxycycline).

C. Patients requiring antibiotic prophylaxis. D. Root surface restorations at the site of recession. E. No detectable CEJ F. Patients who fail to maintain acceptable oral hygiene levels at the test and adjacent teeth.

G. Patients who are pregnant or lactating. H. Patients who use tobacco products (smoking or smokeless tobacco). I. Patients with alcohol abuse problems. J. Patients undergoing long-term steroid therapy. K. History of previous root coverage procedures, graft or GTR, on the test teeth.

L. Patients who fail to complete the informed consent form.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2017-11-30 (Actual); Primary Completion 2018-08-21 (Actual); Study Completion 2018-08-21 (Actual)

PRIMARY OUTCOMES:
Percent root coverage | Six months
  Between 0 and 100%

SECONDARY OUTCOMES:
Creeping Attachment | Six months
  Amount in millimeters

CONTACTS AND LOCATIONS:
Overall Officials: Henry Greenwell, Principal Investigator — University of Louisville
Locations (1):
- Graduate Periodontics, UofL School of Dentistry, Louisville, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No